CLINICAL TRIAL: NCT06748625
Title: Tailored, Multidomain, and Coach-assisted Digital Program for the Adoption and Maintenance of a Healthy Lifestyle in Middle-aged and Older Adults With Modifiable Risk Factors for Dementia: An Efficacy Study
Brief Title: Efficacy of a Multidomain Intervention on Lifestyle Risk Factors for Dementia Prevention
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: LuciLab (Industry)
Collaborators: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other); Sojecci II Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LUCI-03
Record Dates: First submitted 2024-12-18; First posted 2024-12-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Risk Behavior; Cognitive Decline
Keywords: Primary Prevention; Aging; Cognition
MeSH Terms: conditions — Risk-Taking; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luci intervention (Experimental): Participants enrolled in this group will receive the Luci intervention for a 24-week period.
  Interventions: Behavioral: Luci Coach-Assisted Intervention
- Wait-list Control (No Intervention): Participants in the waiting-list control group will not receive any intervention during the study. They will be invited to participate in the program at the end of the trial.

INTERVENTIONS:
Behavioral: Luci Coach-Assisted Intervention — The Luci intervention is a personalized behaviour change program delivered via an interactive web platform with the online support of a coach. It targets 3 lifestyle domains: physical activity, healthy diet and cognitive engagement. Participants will be encouraged to adopt a healthy lifestyle, as a means for cognitive decline/dementia risk reduction. This will be achieved by providing educational materials, practical tips and strategies, and by assisting participants outlining SMART goals to progressively adopt and maintain a healthier lifestyle. Coaching sessions will be held on a weekly basis from week 1 to 12, and every 2 weeks from week 13 to 24.
  Arms: Luci intervention

SUMMARY:
Alzheimer's Disease (AD) and other Dementias have far-reaching consequences on the lives of sufferers and their loved ones, not to mention the impact on the healthcare system. Several studies have identified protective lifestyle habits that might help reduce the risk of cognitive decline: cognitive engagement, physical activity, and a healthy diet. Our aim is to determine the efficacy of the Luci program, an online, coach-assisted, multidomain, behavioural intervention designed to help middle-aged to older adults reduce their risk of dementia by improving their lifestyle habits. In this study, we hope to demonstrate that participating in the Luci program helps to improve lifestyle habits and that the program could therefore become an effective health promotion tool.

DETAILED DESCRIPTION:
Multidomain lifestyle interventions supported by technology might help dementia prevention by reducing the risk associated with lifestyle behaviours. The goal of Luci is to help middle-aged to older adults improve modifiable lifestyle risk factors (diet, physical activity and cognitive engagement) associated with cognitive decline. The intervention is a theory-based, tailored, multidomain, coach-assisted program offered through an interactive online platform promoting healthy lifestyle behaviour changes and their maintenance.

The project deployment follows the Obesity-Related Behavioural Intervention Trials (ORBIT) model. A proof-of-concept study (NCT04616794) was conducted followed by a feasibility study (NCT05141578). All targets (recruitment, enrolment, retention, acceptability, and adherence) were met, which suggests that the protocol is feasible and acceptable and supports moving forward to the efficacy trial.

This study is a 2-arm, randomized, single-blind, parallel-group study aiming to assess the immediate post-intervention (24-weeks) effects of the Luci intervention and their 52-week maintenance, compared to a Waitlist condition in at-risk middle-aged to older individuals. Assessments will be done at Screening (T0), Baseline (T1), week 12 (T2), week 24 (T3), and week 52 (T4).

The primary objective of this study is to determine whether the Luci intervention can result in a greater number of people reducing their behavioural risks when compared to the Waitlist condition. It is hypothesised that the proportion of people with a significant risk reduction will be higher in the Luci condition than in the Waitlist condition.

Individuals assigned to the Intervention group have weekly (weeks 1-12) or bi-monthly (weeks 13-24) sessions with their coach. Coaching sessions last 30 or 60 minutes and are conducted by video call and/or through a chat system.

Throughout the coaching sessions, participants are assisted in creating personalised behavioural SMART (specific, measurable, attainable, relevant and time bound) goals. Coaches also provide motivational support as well as tools to help participants maintain their behaviour changes.

ELIGIBILITY:
Inclusion Criteria :

* Aged between 50 and 75;
* Proficient or native speakers in French or English;
* Computer literate defined as being able to read mails and browse the Internet, and having access to a computer or tablet with an Internet connection;
* Eligible in at least one of the 3 intervention domains, where eligibility is defined as follows:

  * Low cognitive engagement in cognitively stimulating activities, defined as a score ≤ 22 on the adapted Cognitive Activity Questionnaire;
  * Low level of physical activity defined as less than 150 minutes/week) of moderate to vigorous physical activity measured using the Godin- Shephard Leisure Time Physical Activity Questionnaire, and no medical contraindication to physical activity based on the Physical Readiness Questionnaire for Everyone (PAR-Q+);
  * Low adherence to the Mediterranean-type diet defined as a score of ≤ 8 on the adapted Canadian Mediterranean Diet Scale, and no dietary restriction, severe allergy or intolerance or history of eating disorder.

Exclusion Criteria :

* Presence of a cognitive impairment as measured by the Creyos Dementia Assessment;
* General anesthesia within the last 6 months;
* Previous participation in the Luci program or in any validation studies related to the program;
* Current participation in another study;
* Unable to commit participation over the period of the study;
* Being in the precontemplation stage of change;
* High level of perceived stress;
* Having received a diagnosis of :

  * Dementia or neurodegenerative disease (AD and other dementias);
  * Past or present neurological disorder (multiple sclerosis, brain tumour, epilepsy, stroke, traumatic brain injury);
  * Severe psychiatric disorder (schizophrenia, major depression, bipolar disorder);
  * Diabetes or hypertension without medical monitoring;
  * Alcoholism or drug addiction;
  * Any other condition expected to limit participation (e.g., low visual acuity).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Lifestyle Risk Reduction criterion | Change from Screening to Week 24
  The primary endpoint is the number of participants showing a clinically significant change (CSC) from Screening to Week 24 in at least one eligible domain (cognitive engagement, physical activity, mediterranean diet adherence).
Cognitive Engagement | Screening, Week 12, Week 24, Week 52
  Cognitive engagement is measured using the Vemuri Cognitive Activity Questionnaire. Participants are asked to indicate the frequency in which they engage in 10 types of cognitive leisure activities. Scores range from 0 to 70. A higher score represents a higher cognitive engagement level. A clinically significant change is defined as a 6-point minimum increase.
Physical Activity | Screening, Week 12, Week 24, Week 52
  Physical activity is measured using the modified Godin-Shephard Leisure Time Physical Activity Questionnaire which consists of three sets of questions (6 items). An overall physical activity score is computed in Metabolic equivalent tasks (MET)-minutes/week, as well as a moderate-to-vigorous physical activity (MVPA) score. A higher MET value represents a higher physical activity level. A clinically significant change is defined as a 300 MET-min/week minimum increase in the MVPA score.
Mediterranean Diet Adherence | Screening, Week 12, Week 24, Week 52
  Adherence to the Mediterranean Diet is measured with an adaptation of the Canadian Mediterranean Diet Scale. The scale consists of 13 questions on food consumption frequency and intake habits. Scores range from 0 to 13, where a higher score represents a higher adherence level. A clinically significant change is defined as a 2-point minimum increase.

SECONDARY OUTCOMES:
Quality of Life | Baseline, Week 24, Week 52
  Quality of life is measured with the SF-12v2, a 12-item questionnaire.
Cognitive Performance | Screening, Week 24, Week 52
  Cognitive Performance is assessed using the Creyos Dementia Assessment, a computer-administered cognitive test battery that includes 6 tasks measuring 3 cognitive domains (memory, reasoning and verbal abilities). Several scores are calculated: one for each of the 6 individual tests, one for each of the 3 cognitive domains, as well as an overall score. Higher scores indicate higher cognitive performance.

OTHER OUTCOMES:
Multifactorial index of dementia risk | Baseline, Week 24, Week 52
  The CAIDE (Cardiovascular risk factors, aging, and incidence of dementia) is a multifactorial risk estimation scale using age, hypertension, hypercholesterolemia, physical activity level, obesity (BMI), and educational level. A higher score indicates a higher risk of dementia.
Perceived Stress | Screening, Week 24, Week 52
  Perceived stress is investigated using a single question answered on a 5-item Likert scale where a higher score indicates a higher stress level.
Sleep Quality | Baseline, Week 24, Week 52
  Sleep quality is assessed using a single question taken from the Pittsburgh Sleep Quality Index. The score is derived from a 4-point Likert scale where a higher score indicates worse sleep quality.
Anxiety Symptoms | Baseline, Week 24, Week 52
  Anxiety symptoms over the past 2 weeks are assessed using the Generalized Anxiety Disorder (GAD-7) Scale which comprises 7 items which are scored "0" (Not at all) to "3" (Nearly every day) for a maximum total score of 21. A higher score indicates higher anxiety symptoms.
Curent Memory Concerns | Baseline, Week 24, Week 52
  Current memory concerns are evaluated with a single 3-item question.
Readiness to Change | Baseline, Week 12, Week 24, Week 52
  Readiness to change is assessed for each of the 3 intervention domains using a question with five answer options.
Self-efficacy | Baseline, Week 12, Week 24, Week 52
  Self-efficacy is evaluated with the General Self-Efficacy (GSE) Scale which consists of 10 items which are scored from "1" (Not True At All) to "4" (Exactly True) for a maximum score of 40. A higher score indicates greater self-efficacy.
Motivations | Baseline, Week 12, Week 24, Week 52
  Motivations are assessed via the Treatment Self-Regulation Questionnaire (TSRQ), which assesses different forms of motivation. It consists of 15 items, each rated on a 7-point scale ranging from 1 (not at all true) to 7 (very true). The items are combined into 4 subscales, for which 4 subscores can be calculated. Each subscore ranges from 1 to 7, with a higher subscore indicating higher importance of that form of motivation.
Dementia Literacy | Baseline, Week 12, Week 24, Week 52
  Dementia literacy is assessed using 20 questions answered using 5-point Likert scales for a maximum score of 100. A higher score indicates better dementia literacy.
Perceived Progress | Week 12, Week 24, Week 52
  Perceived progress will be measured with one question rated on a 5-point Likert scale for each intervention domain.
Luci Cognitive Engagement Score | Baseline, Week 12, Week 24, Week 52
  In the Luci Cognitive Engagement Questionnaire, 14 types of cognitively stimulating leisure activities are provided, and participants are asked to indicate the frequency in which they engage in those activities. Each question is rated from 0 (Never) to 7 (Every day), for a maximum total score of 98. A higher score represents a higher cognitive engagement level.
Luci Physical Activity Score | Baseline, Week 12, Week 24, Week 52
  In the Luci Physical Activity Questionnaire, participants choose which activities they engage in from a list of almost 70 physical activities. For the selected activities, they are asked to indicate frequency, duration and intensity. Responses are used to calculate the Luci Physical Activity score as well as 3 subscores related to aerobic exercise, muscular resistance, and flexibility training, respectively. A higher score represents a higher physical activity level.
Luci Medi Diet Adherence Score | Baseline, Week 12, Week 24, Week 52
  The Luci Medi Diet Adherence Questionnaire consists of 15 questions on consumption frequency for 13 food groups that are considered characteristic of the Mediterranean diet. A subscore ranging from 0 to 3 is assigned to each food group. Total scores range from 0 to 39, where a higher score represents a higher adherence level.
Health Service Utilisation | Baseline, Week 24, Week 52
  Health care utilisation is assessed using a questionnaire that collects self-reported number of visits to physicians, mental health providers, other providers, emergency department as well as hospital stays, nights in hospital and outpatient surgeries. Total score is the sum of all visits, hospital stays and nights.
Retention Rate | Week 24, Week 52
  Retention rate is the proportion of randomized participants completing at least one of the measures at T3 and T4
Program Adherence | Week 24
  Program adherence is defined as the proportion of participants from the Luci condition who adhered to the program. Participants are considered adherent if they complete at least 12 of the 18 coaching sessions.
Platform Usage | Week 24
  Pattern of use, frequency, duration of use and functionalities used are continuously monitored throughout the program and the data will be analysed.
User Experience | Week 24
  User experience is assessed in participants randomized to the Luci intervention using 36 questions of which 29 are rated on a 5-point Likert scale, 3 are rated on categorical scales, and 4 are free text.
Usability | Week 24
  Usability is assessed using the System Usability Scale (SUS) a five-item questionnaire rated with a 5-point Likert scale.
Goal Attainment | Weekly up to Week 12, then bi-weekly up to Week 24
  Goal attainment and perceived effort to reach the goal are rated by participants in the Luci intervention arm before each coaching sessions. These are reported using 3-point scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucilab, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No